CLINICAL TRIAL: NCT03052244
Title: tDCS Stimulation Combined With VI as a Possible Therapy for Enhancing Functional Ability in SCI With Neuropathic Pain
Brief Title: tDCS and VI to Treat Neuropathic Pain and Function in SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, motti ratmansky, Director, Pain Unit, Loewenstein Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Loe160029CTIL
Record Dates: First submitted 2017-01-29; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: SCI - Spinal Cord Injury
Keywords: tDCS (trans cranial direct current stimulation); Visual illusion; Neuropathic pain; Spinal cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Illusions; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- intervention tDCS+VI (Experimental): The anode will be placed over C3-C4 (EEG 10/20 system) to target M1 and the cathode over the contralateral supraorbital area. The stimulation will apply to the hemisphere which contralateral to the more painful hemi body. 2mA will be delivered over 20 min via neuroConn DC stimulator combined with video presenting walking legs. A total of 10 sessions (5 per week) will be administrated at the same manner.
  Interventions: Device: tDCS+VI
- tDCS Sham+VI Sham (Sham Comparator): The stimulation will be turned on for only short duration (up to 30 sec), the video film will contains graphical illustrations or nature movie without human movement.
  Interventions: Device: tDCS Sham+VI Sham

INTERVENTIONS:
Device: tDCS+VI — 2mA will be delivered over 20min to M1 via neuroConn DC stimulator combined with video presenting walking legs.
  Other Names: transcranial direct current stimulation+visual illusion
  Arms: intervention tDCS+VI
Device: tDCS Sham+VI Sham — 2mA will be delivered up to 30 sec to M1 via neuroConn DC stimulator combined with video presenting graphical illustration or nature movie for total duration of 20 min.
  Other Names: Sham
  Arms: tDCS Sham+VI Sham

SUMMARY:
Transcranial direct current stimulation (tDCS) over the primary motor cortex (M1) will be applied for patient who suffer from neuropathic pain following spinal cord injury The tDCS treatment will be coupled with a video of a man walking (creating a visual illusion) in order to enhance functional ability and reduce pain

DETAILED DESCRIPTION:
Non-invasive cortical brain stimulation is a promising method for treating cases of neuropathic pain in patients with spinal cord injury (SCI). Transcranial direct current stimulation (tDCS) over the primary motor cortex (M1) appears to modulate cortical excitability and can reduce pain levels following SCI, however its effects remaining for short-term and may not be useful for the rehabilitation progress in these patients.

Recent findings suggest that M1 stimulation combined with visual illusion (VI) enhances the reduction in pain which maintain up to 3 month following treatment. The current study aims to reveal whether reduction of neuropathic pain in patients with SCI through tDCS have beneficial effect on functional ability during rehabilitation program.

In the present study the investigators will use anodal stimulation of the M1 via neuroConn DC stimulator. Current intensity of 2mA or sham stimulation will be given during 20 min in parallel to a visual illusion of walking legs (or neutral video for sham stimuli).

ELIGIBILITY:
Inclusion Criteria:

1. patients hospitalized in spinal cord rehabilitation department
2. neuropathic pain following spinal cord injury
3. able to seat on a wheel chair
4. able to understand and comply with basic instructions
5. Hebrew speakers

Exclusion Criteria:

1. epilepsy
2. pregnancy
3. non-neuropathic pain
4. medical condition that affect cognitive functioning
5. medical condition other then the spinal cord injury that affect functioning

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-15 (Estimated); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
change in SCIM 3 (scale) | up to 7 day before and following the treatment
  spinal cord independence measure

SECONDARY OUTCOMES:
change in VAS (Visual Analog Scale) | up to 7 day before and following the treatment
  reported subjective pain scale
change in BPI (Brief Pain Inventory) | up to 24h before and following the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Motti Ratmansky, MD, Principal Investigator — Loewenstein Rehabilitation Center

IPD SHARING:
Plan to Share IPD: No